CLINICAL TRIAL: NCT05557760
Title: Evaluating the Effects of Personalized Booster Sessions on Depression Vulnerability Following Cognitive Control Training for Remitted Depressed Individuals
Brief Title: Effects of Booster Sessions on Depression Vulnerability Following Cognitive Control Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other); Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BC-11832
Record Dates: First submitted 2022-09-21; First posted 2022-09-28 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Major Depression in Remission
Keywords: Depression; Remission; Relapse Prevention; Cognitive Control Training; Internet Intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Control Training Group (Experimental)
  Interventions: Behavioral: Cognitive Control Training (CCT)
- Cognitive Control Training + Booster Sessions Group (Experimental)
  Interventions: Behavioral: Cognitive Control Training (CCT) + Booster Sessions

INTERVENTIONS:
Behavioral: Cognitive Control Training (CCT) — The CCT training group without booster sessions will receive 10 training sessions with the Adaptive Paced Auditory Serial Addition Task (aPASAT). The aPASAT is a Cognitive Control Training where participants need to click on the sum of the last two heard digits.
  Task difficulty is modified based on the participants' current task performance, allowing training of cognitive control.
  Arms: Cognitive Control Training Group
Behavioral: Cognitive Control Training (CCT) + Booster Sessions — The CCT with booster sessions group will receive 10 training sessions with the Adaptive Paced Auditory Serial Addition Task (aPASAT). After these training sessions, participants in this condition will be asked to complete additional CCT sessions after reporting two consecutive assessments of increased depressive symptoms during the monitoring period (PHQ-9 scores equal or greater to 9). Specifically, they will then be instructed to perform three additional sessions within one week. This may be repeated when the participant reports multiple consecutive assessments of increased depressive symptoms during the post-training phase, with a minimum of 3 weeks between the booster sessions and a maximum of 9 boosters (3 x 3 sessions) in total.
  Arms: Cognitive Control Training + Booster Sessions Group

SUMMARY:
The current study aims to examine the impact of booster sessions of cognitive control training (CCT) on indicators of depression vulnerability. Remitted depressed individuals (RMD) will be randomized over two groups, each receiving 10 sessions of the adaptive Paced Auditory Serial Addition Task, a well-established CCT procedure (Koster et al., 2017; Siegle et al., 2007). During and following completion of the training procedure, functioning will be monitored on a weekly basis over a period of 15 weeks. During this period, one group will be offered booster sessions based on early warning signs for possible recurrence of depression, whilst the other group will not receive booster sessions.

DETAILED DESCRIPTION:
Cognitive impairments are closely associated with depression and recent studies have found that these cognitive problems can persist following remission of depression. Internet-delivered cognitive control training (CCT), and the adaptive Paced Auditory Serial Addition Task (aPASAT) in particular, has shown to be an effective preventative intervention for remitted depressed individuals (RMD), where beneficial effects have been found for rumination, depressive symptomatology (Hoorelbeke & Koster, 2017), and risk for recurrence of depression (Hoorelbeke et al., 2021). At the same time, prior studies suggest significant heterogeneity in response to CCT, where RMD individuals can show strong fluctuations in functioning in the months following completion of aPASAT training. In line with this, recent findings suggest that, for individuals with high-risk profiles, initial training gains may diminish over time, resulting in recurrence of internalizing symptomatology (Hoorelbeke et al., 2022). As such, there may be merit in the use of CCT booster sessions.

Currently, it is unclear whether offering additional CCT sessions when RMD individuals are reporting increased symptomatology (i.e., adding booster sessions based on early warning signs for possible recurrence of depression) can increase the long-term effectiveness of CCT. In this study, two groups of RMD individuals will perform 10 CCT sessions, after which one group will be offered booster sessions (contingent on indicators of functioning). For this purpose, we will rely on 15 weekly mobile assessments, using the PHQ-9 questionnaire. In addition, functioning will be assessed using a more extensive assessment battery at baseline, post-training (2 weeks after baseline) and follow-up (15 weeks after baseline).

ELIGIBILITY:
Inclusion Criteria:

* History of ≥ 1 depressive episode(s)
* Currently in remission (≥ 3 months)
* Access to a computer with an internet connection
* Access to a smartphone

Exclusion Criteria:

* Ongoing depressive episode
* Psychotic disorder (current and/or previous)
* Neurological impairments (current and/or previous)
* Excessive substance abuse (current and/or previous)
* Use of antidepressant medication is allowed if kept at a constant level

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9) | weekly assessments from baseline until follow-up (15 weeks after baseline)
  Self-report questionnaire measuring depression symptomatology, with higher scores indicating more severe depression symptoms.

SECONDARY OUTCOMES:
Change in Beck Depression Inventory (BDI-II-NL) | baseline, post training (2 weeks after baseline), follow-up (15 weeks after baseline)
  Self-report questionnaire measuring depression symptomatology, with higher scores indicating more severe depression symptoms.
Change in Perseverative Thinking Questionnaire (PTQ-NL) | baseline, post training (2 weeks after baseline), follow-up (15 weeks after baseline)
  Change from baseline in repetitive negative thinking. The PTQ-NL consist of 15 items which are rated from 0 (never) to 4 (almost always). Lower scores indicate lower levels of repetitive negative thinking.
Change in Cognitive Emotion Regulation Questionnaire (CERQ) | baseline, post training (2 weeks after baseline), follow-up (15 weeks after baseline)
  Self-report measure for emotion regulation: a 36-item questionnaire, consisting of adaptive and maladaptive emotion regulation strategies. Each item is rated on a 1 to 5 scale (1 = almost never and 5 = almost always).
Change in Adult Temperament Questionnaire (ATQ), Effortful Control subscale | baseline, post training (2 weeks after baseline), follow-up (15 weeks after baseline)
  Measured by the subscale Effortful Control (EC) from the Adult Temperament Questionnaire (ATQ).
Change in Burnout Assessment Tool (BAT) | baseline, post training (2 weeks after baseline), follow-up (15 weeks after baseline)
  The Burnout Assessment Tool (BAT) is used to assess burn-out risk. The score ranges from 1 to 5, with higher scores indicating a higher risk of burn-out
Change in Remission from Depression Questionnaire (RDQ-NL) | baseline, post training (2 weeks after baseline), follow-up (15 weeks after baseline)
  The Remission from Depression Questionnaire has 41 items, which assess domains such as positive mental health, life satisfaction, and sense of well-being. The items are scored 0 (not at all or rarely true), 1 (sometimes true) or 2 (often or almost always true).
Change in non-adaptive PASAT performance | baseline, post training (2 weeks after baseline), follow-up (15 weeks after baseline)
  A non-adaptive computerized version of the Paced Auditory Serial- Addition Task (PASAT) was used as a measure of participants' working memory abilities. Higher accuracy scores suggest greater cognitive control resources.
Change in Work Productivity and Activity Impairment Questionnaire (WPAI) | baseline, follow-up (15 weeks after baseline)
  The 6-item WPAI measures the effect of health problems on the ability to work and carry out daily activities.
Change in Short Form Health Survey (SF-36) | baseline, follow-up (15 weeks after baseline)
  The 11-item SF-36 measures attitudes on general health.
Change in questionnaire based on the Medical Consumption Questionnaire (iMCQ) | baseline, follow-up (15 weeks after baseline)
  The iMCQ measures healthcare consumption.

OTHER OUTCOMES:
Change in List of Threatening Experiences (LTE-Q) | baseline, post training (2 weeks after baseline), follow-up (15 weeks after baseline)
  In the LTE questionnaire, unpleasant life events are listed and participants are asked if these events occurred recently. The LTE-Q contains 13 items for which "yes" or "no" are the two possible answers. This questionnaire is included to be able to check for occurrence of life events during the intervention- and follow-up period.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Ghent, Oost-Vlaanderen
  - Ghent University, Ghent, Oost-Vlaanderen

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized individual participant data can be stored on Open-Science Framework (OSF).
Supporting Information: Analytic Code